CLINICAL TRIAL: NCT05106114
Title: Intensive Gait Training Rehabilitation Protocol to Enhance Functional Parameters of Walking After Single-event Multi-level Surgery in Cerebral Palsy
Brief Title: Intensive Gait Training Rehabilitation Protocol After Surgery in Cerebral Palsy
Acronym: ACTIV'MARCHE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondation Ellen Poidatz (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RIRCM-P2021-1
Record Dates: First submitted 2021-05-28; First posted 2021-11-03 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intensive gait training rehabilitation protocole (Experimental): * Functional gait training
  * Strengthening interventions
  * High intensity interval training
  Interventions: Other: Intensive gait training rehabilitation protocole

INTERVENTIONS:
Other: Intensive gait training rehabilitation protocole — 6 weeks of intensive gait training : 4 weeks at the center and 2 weeks of home-based telerehabilitation

SUMMARY:
In the context of cerebral palsy, rehabilitation post Single-Event Multi-Level Surgery (SEMLS) is a long process. One year after surgery and rehabilitation, the functional benefits are usually less improved than the gait pattern. This may be caused by a lack of intensity in the final rehabilitation steps. Thus we created an intensive gait training rehabilitation protocole. This protocole associates 4 weeks of intensive rehabilitation in a healthcare center followed by 2 weeks of intensive rehabilitation at home. The objective of this study is to evaluate the efficiency of this protocol to improve walking speed and endurance, gross motor function et muscular strength.

ELIGIBILITY:
Inclusion Criteria:

* Cerebral palsy
* Age between 10 and 20 years
* Single-Event multi-level surgery more than one year ago
* GMFCS I to III
* Capacity to understand simple instructions
* Volontary consent

Exclusion Criteria:

* injuries or pain in lower limbs
* toxines or surgery less than one year before the study

Ages: 10 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 23 (Actual)
Dates: Start 2021-05-28 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-05-30 (Actual)

PRIMARY OUTCOMES:
6-minutes walking test | 15 minutes
  Evaluation of walking speed

SECONDARY OUTCOMES:
Gross Motor Function Measure (GMFM) | 30 minutes
  Evaluation of Gross motor function
10 meters walking test | 5 minutes
  Evaluation of walking speed
Shuttle Run test-I and II | 10 minutes
  Evaluation of aerobic capacity
Muscle strength via a Dynamometer | 15 minutes
  Evaluation of muscle strength
Spatio-temporal gait parameters | 45 minutes
  Cadence, Walking speed, Step Length,Step Time,Step Width
Number of steps per day | one week wearing an accelerometer
Pediatric Quality of Life Inventory (PedSQL) | 10 minutes
  Evaluation of quality of life via a questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Michel Bams, MD, Principal Investigator — Medical Doctor; Eric Desailly, PhD, Study Director — Director of research
Locations (1):
- Fondation Ellen Poidatz, Saint-Fargeau-Ponthierry, France

IPD SHARING:
Plan to Share IPD: No